CLINICAL TRIAL: NCT01889186
Title: A Phase 2 Open-Label Study of the Efficacy of ABT-199 (GDC-0199) in Subjects With Relapsed/Refractory or Previously Untreated Chronic Lymphocytic Leukemia Harboring the 17p Deletion
Brief Title: A Study of the Efficacy of ABT-199 in Subjects With Relapsed/Refractory or Previously Untreated Chronic Lymphocytic Leukemia With the 17p Deletion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M13-982; 2012-004027-20 (EudraCT Number)
Expanded Access: NCT03123029 (Available)
Record Dates: First submitted 2013-06-26; First posted 2013-06-28 (Estimated); Results first posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-11

CONDITIONS: Chronic Lymphocytic Leukemia; 17p Deletion; Cancer of the Blood and Bone Marrow
Keywords: Chronic Lymphocytic Leukemia; 17p Deletion
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Chromosome 17 deletion | interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Main Cohort (Experimental): Participants received ABT-199 tablets once daily (QD) orally for up to 79 months. The starting dose was 20 mg daily, increasing over a period of 5 weeks up to the daily dose of 400 mg.
  Interventions: Drug: ABT-199 (Main Cohort)
- Safety Expansion Cohort (Experimental): Participants received ABT-199 tablets once daily (QD) orally for up to 68 months. The starting dose was 20 mg daily, increasing over a period of 5 weeks up to the daily dose of 400 mg.
  Interventions: Drug: ABT-199 (Safety Expansion Cohort)

INTERVENTIONS:
Drug: ABT-199 (Main Cohort) — Participants received a test dose of ABT-199 of ≤ 20 mg on Week 1 Day 1 of the Lead-In Period. For those with significant electrolyte and/or lymphocyte changes within 24 hours of the first dose, the 20 mg dose was maintained for 7 days with escalation to 50 mg on Week 2 Day 1. If none of the electrolyte and/or lymphocyte changes occurred within 24 hours from ABT-199 20 mg dose administration, the participant was dose-escalated to 50 mg on Week 1 Day 2. After the first dose of 50 mg, if no laboratory abnormalities occurred, the participant remained on the 50 mg dose through Week 1. After receiving the 50 mg dose for approximately 1 week (6 to 7 days), the following dose escalation proceeded with weekly increases in dose: → 100 mg → 200 mg → 400 mg (or additional lead-in steps to designated 400 mg dose), as tolerated.
  Other Names: Venetoclax; GDC-0199
  Arms: Main Cohort
Drug: ABT-199 (Safety Expansion Cohort) — Participants received an initial dose of ABT-199 of 20 mg on Week 1 Day 1 of the Lead-In Period. If one or more electrolyte changes (from the 0 hr measurement prior to dosing) suggestive of laboratory tumor lysis syndrome (LTLS) or clinical TLS (CTLS) occurred within 24 hours of the 20 mg dose, no additional doses were administered until resolution. Upon resolution of laboratory abnormalities, the 20 mg dose was continued through Week 1. If no significant findings suggestive of clinical or laboratory TLS occurred within 24 hours, the 20 mg dose was continued through Week 1 Day 7, and escalated to a dose of 50 mg on Week 2 Day 1. Those who had drug interruptions may have been allowed to escalate to and be maintained at 50 mg for 1 week after they had been on a 20 mg dose for at least 1 week (5 - 7 days). After a week at 50 mg, weekly dose escalations were implemented as follows: 100 mg → 200 mg → 400 mg (or additional lead-in steps to designated 400 mg dose) as tolerated.
  Other Names: Venetoclax; GDC-0199
  Arms: Safety Expansion Cohort

SUMMARY:
This was an open-label, multicenter, global study to determine the efficacy of ABT-199 (Venetoclax) monotherapy in participants with relapsed/refractory (R/R) or previously untreated chronic lymphocytic leukemia (CLL) harboring 17p deletion.

DETAILED DESCRIPTION:
This study was designed to enroll approximately 150 participants in 2 cohorts: a main cohort of approximately 100 participants, and a safety expansion (SE) cohort of approximately 50 participants. The primary objective of the main cohort was to evaluate the efficacy of ABT-199 monotherapy in participants with R/R CLL harboring the 17p deletion. The primary objective of the safety expansion cohort was to evaluate the safety of ABT-199 in approximately 50 participants with R/R CLL harboring 17p deletion treated per updated tumor lysis syndrome (TLS) prophylaxis and management measures.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be greater than or equal to 18 years of age.
* Participant must have diagnosis of chronic lymphocytic leukemia (CLL) that meets published 2008 Modified IWCLL NCI-WG (International Workshop for Chronic Lymphocytic Leukemia National Cancer Institute-Working Group) Guidelines.

  * Participant has an indication for treatment according to the 2008 Modified IWCLL NCI WG Guidelines;
  * Participant has clinically measurable disease (lymphocytosis > 5 × 10^9/L and/or palpable and measurable nodes by physical exam and/or organomegaly assessed by physical exam);
  * Participant must be refractory or have relapsed after receiving at least one prior line of therapy (participants that have progressed after 1 cycle of treatment or have completed at least 2 cycles of treatment for a given line of therapy) or previously untreated CLL (previously untreated CLL participants must have received no prior chemotherapy or immunotherapy. Participants with a history of emergency, loco-regional radiotherapy (e.g., for relief of compressive signs or symptoms) are eligible. In addition, participants must meet the CLL diagnostic criteria above and must have > 5 × 10^9/L B-Lymphocytes in the peripheral blood.);
  * Participants must have 17p deletion, assessed by local laboratory (in bone marrow or peripheral blood) or assessed by central laboratory (peripheral blood).
* Participant has an Eastern Cooperative Oncology Group (ECOG) performance score of less than or equal to 2.
* Participant must have adequate bone marrow function at Screening as follows:

  * Absolute Neutrophil Count (ANC) greater than or equal to 1000/µL, or
  * For subjects with an ANC less than 1000/µL at Screening and bone marrow heavily infiltrated with underlying disease (unless cytopenia is clearly due to marrow involvement of CLL), growth factor support may be administered after Screening and prior to the first dose of ABT-199 to achieve the ANC eligibility criteria (greater than or equal to 1000/µL);
  * Platelets greater than 30,000/mm^3 (without transfusion support within 14 days of Screening, without evidence of mucosal bleeding, without known history of bleeding episode within 3 months of Screening, and without history of bleeding disorder);
  * Hemoglobin greater than or equal to 8.0 g/dL.
* Participant must have adequate coagulation, renal, and hepatic function, per laboratory reference range at Screening as follows:

  * Activated partial thromboplastin time (aPTT) and prothrombin time (PT) not to exceed 1.5 × the upper limit of normal;
  * Calculated creatinine clearance greater than 50 mL/min using 24-hour Creatinine Clearance or modified Cockcroft-Gault equation (using Ideal Body Mass [IBM] instead of Mass). For participants that have body mass index (BMI) of > 30 kg/m^2 or < 19 kg/m^2, 24-hour measured urine creatinine clearance is required;
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 3.0 × the upper normal limit of institution's normal range; Bilirubin less than or equal to 1.5 × upper limit of normal. Participants with Gilbert's Syndrome may have a bilirubin greater 1.5 × upper limit of normal, per correspondence between the investigator and AbbVie medical monitor.
* For participants at high risk of tumor lysis syndrome a pre-approval by the AbbVie medical monitor is required prior to enrollment.

Exclusion Criteria:

* Participant has undergone an allogeneic stem cell transplant.
* Participant has developed Richter's transformation confirmed by biopsy.
* Participant has prolymphocytic leukemia.
* Participant has active and uncontrolled autoimmune cytopenias (for 2 weeks prior to Screening), including autoimmune hemolytic anemia and idiopathic thrombocytopenic purpura despite low dose corticosteroids.
* Participant has previously received ABT-199.
* Participant has received a biologic agent for anti-neoplastic intent within 30 days prior to the first dose of study drug.
* Participant has received any of the following within 14 days or 5 half-lives as applicable prior to the first dose of study drug, or has not recovered to less than Common Toxicity Criteria (CTC) grade 2 clinically significant adverse effect(s)/toxicity(s) of the previous therapy:

  * Any anti-cancer therapy including chemotherapy, or radiotherapy;
  * Investigational therapy, including targeted small molecule agents.
* Participant has known allergy to both xanthine oxidase inhibitors and rasburicase.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2013-06-27 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2020-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (48):
- United States (16):
  - University of Arizona Cancer Center - North Campus /ID# 96748, Tucson, Arizona
  - City of Hope /ID# 112875, Duarte, California
  - Moore UC San Diego Cancer Center /ID# 91793, La Jolla, California
  - Stanford University School of Med /ID# 105117, Stanford, California
  - Georgetown University Hospital /ID# 96954, Washington D.C., District of Columbia
  - Northwestern University Feinberg School of Medicine /ID# 92499, Chicago, Illinois
  - The University of Chicago Medical Center /ID# 96960, Chicago, Illinois
  - Ingalls Memorial Hosp /ID# 92497, Harvey, Illinois
  - Dana-Farber Cancer Institute /ID# 92494, Boston, Massachusetts
  - Henry Ford Health System /ID# 97795, Detroit, Michigan
  - Hackensack Univ Med Ctr /ID# 92500, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey /ID# 92513, New Brunswick, New Jersey
  - Columbia Univ Medical Center /ID# 103835, New York, New York
  - Columbia Univ Medical Center /ID# 94716, New York, New York
  - Cleveland Clinic Main Campus /ID# 92495, Cleveland, Ohio
  - University of Texas MD Anderson Cancer Center /ID# 92521, Houston, Texas
- Australia (4):
  - Royal North Shore Hospital /ID# 98836, St Leonards, New South Wales
  - John Fawkner Private Hospital /ID# 98835, Coburg, Victoria
  - Peter MacCallum Cancer Ctr /ID# 91795, Melbourne, Victoria
  - Royal Melbourne Hospital /ID# 91794, Parkville, Victoria
- Duplicate_Jewish General Hospital /ID# 99476, Montreal, Quebec, Canada
- France (4):
  - Centre Hospitalier Lyon Sud /ID# 98839, Pierre-Bénite, Auvergne-Rhône-Alpes
  - Hopital Pitie Salpetriere /ID# 98842, Paris
  - Centre Henri Becquerel /ID# 98838, Rouen
  - Hopital Avicenne - APHP /ID# 98840, Bobigny, Île-de-France Region
- Germany (9):
  - Universitaetsklinik Heidelberg /ID# 98845, Heidelberg, Baden-Wurttemberg
  - Uniklinik Koeln /ID# 98847, Cologne, North Rhine-Westphalia
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel /ID# 113235, Kiel, Schleswig-Holstein
  - Universitaetsklinikum Ulm /ID# 92533, Ulm, Thuringia
  - Universitaetsklinikum Carl Gustav Carus an der TU Dresden /ID# 113256, Dresden
  - Universitaetsklinikum Freiburg /ID# 113276, Freiburg im Breisgau
  - Universitaetsmedizin Goettingen /ID# 113258, Göttingen
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz /ID# 113236, Mainz
  - Muenchen Klinik Schwabing /ID# 113275, München
- Poland (3):
  - SP ZOZ Szpital Uniwersytecki w Krakowie /ID# 98849, Krakow, Lesser Poland Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 w Lublinie /ID# 98848, Lublin, Lublin Voivodeship
  - Szpital Wojewodzki w Opolu /ID# 102855, Opole, Opole Voivodeship
- United Kingdom (11):
  - Leicester Royal Infirmary /ID# 98865, Leicester, England
  - The Royal Bournemouth Hospital /ID# 118975, Bournemouth
  - Addenbrookes Hospital /ID# 119977, Cambridge
  - St. James University Hospital /ID# 98863, Leeds
  - Royal Liverpool and Broadgreen /ID# 98860, Liverpool
  - St Bartholomew's Hospital, Bar /ID# 98862, London
  - King's College Hospital NHS Foundation Trust /ID# 119975, London
  - The Christie Hospital /ID# 98864, Manchester
  - Oxford Univ Hosp NHS Trust /ID# 119976, Oxford
  - Derriford Hospital /ID# 118335, Plymouth
  - Royal Marsden Hospital /ID# 98861, Sutton

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Background] Stilgenbauer S, Eichhorst B, Schetelig J, Coutre S, Seymour JF, Munir T, Puvvada SD, Wendtner CM, Roberts AW, Jurczak W, Mulligan SP, Bottcher S, Mobasher M, Zhu M, Desai M, Chyla B, Verdugo M, Enschede SH, Cerri E, Humerickhouse R, Gordon G, Hallek M, Wierda WG. Venetoclax in relapsed or refractory chronic lymphocytic leukaemia with 17p deletion: a multicentre, open-label, phase 2 study. Lancet Oncol. 2016 Jun;17(6):768-778. doi: 10.1016/S1470-2045(16)30019-5. Epub 2016 May 10. PMID 27178240
- [Derived] Stilgenbauer S, Tausch E, Roberts AW, Davids MS, Eichhorst B, Hallek M, Hillmen P, Schneider C, Schetelig J, Bottcher S, Kater AP, Jiang Y, Boyer M, Popovic R, Ghanim MT, Moran M, Sinai WJ, Wang X, Mukherjee N, Chyla B, Wierda WG, Seymour JF. Six-year follow-up and subgroup analyses of a phase 2 trial of venetoclax for del(17p) chronic lymphocytic leukemia. Blood Adv. 2024 Apr 23;8(8):1992-2004. doi: 10.1182/bloodadvances.2023011741. PMID 38290108
- [Derived] Roberts AW, Ma S, Kipps TJ, Coutre SE, Davids MS, Eichhorst B, Hallek M, Byrd JC, Humphrey K, Zhou L, Chyla B, Nielsen J, Potluri J, Kim SY, Verdugo M, Stilgenbauer S, Wierda WG, Seymour JF. Efficacy of venetoclax in relapsed chronic lymphocytic leukemia is influenced by disease and response variables. Blood. 2019 Jul 11;134(2):111-122. doi: 10.1182/blood.2018882555. Epub 2019 Apr 25. PMID 31023700
- [Derived] Stilgenbauer S, Eichhorst B, Schetelig J, Hillmen P, Seymour JF, Coutre S, Jurczak W, Mulligan SP, Schuh A, Assouline S, Wendtner CM, Roberts AW, Davids MS, Bloehdorn J, Munir T, Bottcher S, Zhou L, Salem AH, Desai M, Chyla B, Arzt J, Kim SY, Verdugo M, Gordon G, Hallek M, Wierda WG. Venetoclax for Patients With Chronic Lymphocytic Leukemia With 17p Deletion: Results From the Full Population of a Phase II Pivotal Trial. J Clin Oncol. 2018 Jul 1;36(19):1973-1980. doi: 10.1200/JCO.2017.76.6840. Epub 2018 May 1. PMID 29715056

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All treated participants: all participants who received at least one dose of ABT-199 in either the Main Cohort or Safety Expansion Cohort
Period: Overall Study
Arm/Group | Main Cohort | Safety Expansion Cohort
Started | 107 | 51
Completed | 0 | 0
Not Completed | 107 | 51
Not completed — Adverse event- not related to progression | 18 | 5
Not completed — Adverse event- related to progression | 7 | 2
Not completed — COVID-19 logistical restrictions | 1 | 0
Not completed — Investigator request | 1 | 1
Not completed — Progressive disease- Richter's | 12 | 7
Not completed — Progressive disease per protocol | 46 | 17
Not completed — Stem cell transplant | 2 | 1
Not completed — Withdrew consent | 2 | 3
Not completed — Other, not specified | 18 | 15

BASELINE CHARACTERISTICS:
Population: All treated participants: all participants who received at least one dose of ABT-199 in either the Main Cohort or Safety Expansion Cohort
Groups:
- Total: Total of all reporting groups
Arm/Group | Main Cohort | Safety Expansion Cohort | Total
Number analyzed (Participants) | 107 | 51 | 158
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (9.87) | 65.4 (9.97) | 65.6 (9.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 22 | 59
  Male | 70 | 29 | 99
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 103 | 49 | 152
  Black | 3 | 1 | 4
  Asian | 0 | 0 | 0
  American Indian/Alaska Native | 0 | 0 | 0
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  Other | 0 | 0 | 0
  Multi race | 0 | 0 | 0
  MISSING | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (Main Cohort)
Description: The overall response rate (ORR) is defined as the proportion of participants with an overall response (complete remission [CR] + complete remission with incomplete marrow recovery [CRi] + nodular partial remission [nPR] + partial remission [PR]) per the 2008 Modified International Workshop for Chronic Lymphocytic Leukemia (IWCLL)/National Cancer Institute-Working Group (NCI-CWG) criteria as assessed by the Independent Review Committee (IRC) in the first 70 participants treated in the Main Cohort.
Time Frame: Up to 36 weeks
Population: The first 70 participants who were treated with ABT-199 in the Main Cohort
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Main Cohort
Number analyzed (Participants) | 70
percentage of participants | 77.1 [65.6 to 86.3]
Statistical Analysis 1: Comparison: Main Cohort; The ORR for ABT-199 was tested to reject the null hypothesis of ORR = 40%. If the null hypothesis is rejected and the ORR is higher than 40%, then ABT-199 has been shown to have an ORR significantly higher than 40%.The p-value is from the exact binomial distribution comparing ABT-199 ORR to the 40% historical control rate; Test type: Superiority; p < 0.001, Clopper-Pearson exact method

2. Primary Outcome: Number of Participants With Adverse Events (Safety Expansion Cohort)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study drug. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent adverse events/treatment-emergent serious adverse events (TEAEs/TESAEs) are defined as any event that began or worsened in severity on or after the first dose of study drug.
Time Frame: From the first dose of study drug until 30 days following last dose of study drug (up to 69 months)
Population: All treated participants in the Safety Expansion Cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Expansion Cohort
Number analyzed (Participants) | 51
Participants | 51

3. Secondary Outcome: Overall Response Rate (ORR) (Safety Expansion Cohort)
Description: The overall response rate (ORR) is defined as the proportion of participants with an overall response (complete remission [CR] + complete remission with incomplete marrow recovery [CRi] + nodular partial remission [nPR] + partial remission [PR]) per the 2008 Modified International Workshop for Chronic Lymphocytic Leukemia (IWCLL)/National Cancer Institute-Working Group (NCI-CWG) criteria.
Time Frame: Up to the data cutoff date of 15 June 2017, approximately 4 years of follow-up
Population: All treated participants in the Safety Expansion Cohort
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Safety Expansion Cohort
Number analyzed (Participants) | 51
percentage of participants | 82.4 [69.1 to 91.6]

4. Secondary Outcome: Complete Remission (CR) Rate
Description: Complete remission was defined as the proportion of participants who achieved a CR or Complete Remission with Incomplete Marrow Recovery(CRi ) per the 2008 Modified International Workshop for Chronic Lymphocytic Leukemia (IWCLL)/National Cancer Institute-Working Group (NCI-CWG) criteria. Participants who did not achieve a CR or CRi were considered to be non-responders in the calculation of CR rate.
Time Frame: Up to the data cutoff date of 15 June 2017, approximately 4 years of follow-up
Population: All treated participants in the Main Cohort and the Safety Expansion Cohort
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Main Cohort | Safety Expansion Cohort
Number analyzed (Participants) | 107 | 51
percentage of participants | 21.5 [14.1 to 30.5] | 27.5 [15.9 to 41.7]

5. Secondary Outcome: Partial Remission (PR) Rate
Description: PR rate was defined as the proportion of participants who achieved a nodular partial remission (nPR) or PR per the 2008 Modified International Workshop for Chronic Lymphocytic Leukemia (IWCLL)/National Cancer Institute-Working Group (NCI-CWG) criteria. Participants who did not achieve a nPR or PR were considered to be non-responders in the calculation of PR rate.
Time Frame: Up to the data cutoff date of 15 June 2017, approximately 4 years of follow-up
Population: All treated participants in the Main Cohort and the Safety Expansion Cohort
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Main Cohort | Safety Expansion Cohort
Number analyzed (Participants) | 107 | 51
percentage of participants | 53.3 [43.4 to 63.0] | 54.9 [40.3 to 68.9]

6. Secondary Outcome: Duration of Overall Response
Description: Duration of overall response (DoR) was defined as the number of days from the date of first response (CR, CRi, nPR, or PR) by either CT scan or physical exam determination to the earliest recurrence (progressive disease; PD) or death. For participants who had a PR before CR, CRi, or nPR in subsequent visits, the DoR was computed from the earliest PR. If a participant was still responding, then their data was censored at the date of their last available disease assessment. To be included in the DoR analysis, participants must have had a response per the 2008 Modified International Workshop for Chronic Lymphocytic Leukemia (IWCLL)/National Cancer Institute-Working Group (NCI-CWG) criteria (CR, CRi, confirmed nPR, or confirmed PR). For participants who never experienced response, their data was not included in the analysis.
Time Frame: Up to the data cutoff date of 15 June 2017, approximately 4 years of follow-up
Population: All treated participants in the Main Cohort and the Safety Expansion Cohort with a response and available data
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Main Cohort | Safety Expansion Cohort
Number analyzed (Participants) | 80 | 42
months | 35.3 [26.5 to NA] — Not calculable/estimable due to insufficient number of events | NA [27.3 to NA] — Not calculable/estimable due to insufficient number of events

7. Secondary Outcome: Progression-free Survival
Description: Duration of progression-free survival (PFS) was defined as the number of days from the date of first dose to the date of earliest disease progression or death. All disease progression was included regardless of whether the event occurred while the participant was taking ABT-199 or had previously discontinued ABT-199. If the participant does not experience disease progression or death, then the data was censored at the date of last disease assessment. Data for participants without any disease assessments performed after the baseline visit were censored at the date of first dose plus 1 day.
Time Frame: Up to the data cutoff date of 15 June 2017, approximately 4 years of follow-up
Population: All treated participants in the Main Cohort and the Safety Expansion Cohort with available data
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Main Cohort | Safety Expansion Cohort
Number analyzed (Participants) | 107 | 51
months | 24.7 [21.7 to 35.9] | 30.2 [24.7 to NA] — Not calculable/estimable due to insufficient number of events

8. Secondary Outcome: Event-free Survival
Description: Event-free survival (EFS) was defined as the number of days from the date of first dose to the date of earliest disease progression, death, or start of a new anti-leukemic therapy. If the specified event (disease progression, death, start of a new anti-leukemic treatment) did not occur, participants were censored at the date of last disease assessment. Data for participants without any disease assessments performed after the baseline visit were censored at the date of first dose plus 1 day.
Time Frame: Up to the data cutoff date of 15 June 2017, approximately 4 years of follow-up
Population: All treated participants in the Main Cohort and the Safety Expansion Cohort with available data
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Main Cohort | Safety Expansion Cohort
Number analyzed (Participants) | 107 | 51
months | 24.7 [19.7 to 35.9] | 30.2 [24.7 to NA] — Not calculable/estimable due to insufficient number of events

9. Secondary Outcome: Time to Progression
Description: Time to progression (TTP) was defined as the number of days from the date of first dose to the date of earliest disease progression. All disease progression was included regardless of whether the event occurred while the participant was taking ABT-199 or had previously discontinued ABT-199. If the participant did not experience disease progression, then the data was censored at the date of last available disease assessment. Data for participants without any disease assessments performed after the baseline visit were censored at the date of first dose plus 1 day.
Time Frame: Up to the data cutoff date of 15 June 2017, approximately 4 years of follow-up
Population: All treated participants in the Main Cohort and the Safety Expansion Cohort with available data
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Main Cohort | Safety Expansion Cohort
Number analyzed (Participants) | 107 | 51
months | 28.2 [21.9 to 39.0] | 30.2 [27.0 to NA] — Not calculable/estimable due to insufficient number of events

10. Secondary Outcome: Time to First Response
Description: Time to first response was defined as the number of days from the date of first dose to the date of the first sign of response (CR, CRi, nPR, or PR) given the participant has had a CR, CRi, confirmed nPR, or confirmed PR per the 2008 Modified International Workshop for Chronic Lymphocytic Leukemia (IWCLL)/National Cancer Institute-Working Group (NCI-CWG) criteria. The first response could have been an assessment by physical exam as long as the results were later confirmed per the 2008 Modified IWCLL NCI-WG criteria. For participants who never experienced a response, the participant's data were not included in the analysis.
Time Frame: Up to the data cutoff date of 15 June 2017, approximately 4 years of follow-up
Population: All treated participants in the Main Cohort and the Safety Expansion Cohort with a response and available data
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Main Cohort | Safety Expansion Cohort
Number analyzed (Participants) | 80 | 42
months | 1.1 [1.0 to 1.3] | 1.3 [1.1 to 1.5]

11. Secondary Outcome: Time to 50% Reduction in Absolute Lymphocyte Count
Description: Time to 50% reduction in absolute lymphocyte count (ALC) was defined as the number of days (hours if applicable) from the date of first dose to the date when the ALC had reduced to 50% of the baseline value. Only participants with a baseline of ALC > 5 × 10^9 /L were included in the analysis. For participants who never achieved a 50% reduction in ALC, the participant's data were not included in the analysis.
Time Frame: Up to the data cutoff date of 15 June 2017, approximately 4 years of follow-up
Population: All treated participants with a baseline of ALC > 5 × 10^9 /L, a 50% reduction in ALC, and available data
Measure: Mean (95% Confidence Interval); unit: weeks
Groups:
- All Treated Participants: Participants in the Main Cohort received ABT-199 tablets once daily (QD) orally for up to 79 months,and those in the Safety Expansion Cohort received ABT-199 tablets once daily (QD) orally for up to 68 months. For both groups, the starting dose was 20 mg daily, increasing over a period of 5 weeks up to the daily dose of 400 mg.
Arm/Group | Main Cohort | All Treated Participants
Number analyzed (Participants) | 85 | 125
weeks | 1.1 [0.9 to 1.2] | 1.2 [1.1 to 1.4]

12. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was defined as number of days from the date of first dose to the date of death. For participants who did not die, their data was censored at the date of last study visit or the last known date to be alive, whichever was later.
Time Frame: Up to the data cutoff date of 15 December 2020, approximately 7.5 years of follow-up
Population: All treated participants with available data
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Main Cohort | Safety Expansion Cohort
Number analyzed (Participants) | 107 | 51
months | 53.4 [37.0 to 73.0] | NA [61.6 to NA] — Not calculable/estimable due to insufficient number of events

13. Secondary Outcome: Percentage of Participants Who Moved on to Stem Cell Transplant
Description: The percentage of participants who moved on to stem cell transplant was summarized.
Time Frame: Up to the data cutoff date of 15 June 2017, approximately 4 years of follow-up
Population: All treated participants with available data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Main Cohort | All Treated Participants
Number analyzed (Participants) | 107 | 158
percentage of participants | 2.8 [0.6 to 8.0] | 2.5 [0.7 to 6.4]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the first dose of study drug until 30 days after last study drug administration, up to 80 months for the Main Cohort and up to 69 months for the Safety Expansion Cohort.
Description: TEAEs and SAEs are defined as any AE or SAE with onset or worsening reported by a participant from the time that the first dose of study drug is administered until 30 days have elapsed following discontinuation of study drug. TEAEs were collected whether elicited or spontaneously reported by the participant.
Arm/Group | Main Cohort | Safety Expansion Cohort
All-Cause Mortality (participants affected / at risk) | 62/107 | 19/51
Serious Adverse Events (participants affected / at risk) | 78/107 | 34/51
Other Adverse Events (participants affected / at risk) | 103/107 | 50/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Cohort (N=107) | Safety Expansion Cohort (N=51)
ANAEMIA (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
AUTOIMMUNE HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 7 (10) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 7 (9) | 2 (2)
HAEMOLYSIS (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
HAEMORRHAGIC DIATHESIS (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
IMMUNE THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 (0) | 1 (1)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 1 (1)
ANGINA PECTORIS (Cardiac disorders) | 2 (2) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 3 (3) | 0 (0)
ATRIAL FLUTTER (Cardiac disorders) | 1 (1) | 0 (0)
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 1 (1)
CARDIOGENIC SHOCK (Cardiac disorders) | 1 (1) | 0 (0)
CARDIOPULMONARY FAILURE (Cardiac disorders) | 2 (2) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 2 (3) | 0 (0)
HYPERTENSIVE HEART DISEASE (Cardiac disorders) | 1 (1) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 2 (2)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 (1) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
ATRIAL SEPTAL DEFECT (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
HYDROCELE (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
RETINAL ARTERY OCCLUSION (Eye disorders) | 1 (1) | 0 (0)
VISION BLURRED (Eye disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 (2) | 0 (0)
APHTHOUS ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
ASCITES (Gastrointestinal disorders) | 1 (1) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 2 (2)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
ENTERITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
INTESTINAL PSEUDO-OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
TOOTH LOSS (Gastrointestinal disorders) | 1 (1) | 0 (0)
UMBILICAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 (2) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 1 (1)
GAIT DISTURBANCE (General disorders) | 1 (1) | 0 (0)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 4 (4) | 1 (1)
HYPOTHERMIA (General disorders) | 1 (1) | 0 (0)
IMPAIRED HEALING (General disorders) | 1 (1) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 2 (2) | 0 (0)
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 1 (1) | 0 (0)
PAIN (General disorders) | 1 (1) | 0 (0)
PERFORMANCE STATUS DECREASED (General disorders) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 8 (8) | 0 (0)
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 1 (1) | 0 (0)
CHOLANGITIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 1 (1) | 0 (0)
HYPOGAMMAGLOBULINAEMIA (Immune system disorders) | 0 (0) | 1 (1)
ADENOVIRUS INFECTION (Infections and infestations) | 1 (1) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 1 (1)
BETA HAEMOLYTIC STREPTOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
BRONCHITIS (Infections and infestations) | 2 (2) | 0 (0)
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 1 (1) | 0 (0)
CAMPYLOBACTER INFECTION (Infections and infestations) | 1 (2) | 0 (0)
CELLULITIS (Infections and infestations) | 2 (2) | 0 (0)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 (2) | 0 (0)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 2 (3) | 0 (0)
EMPYEMA (Infections and infestations) | 0 (0) | 1 (1)
ERYSIPELAS (Infections and infestations) | 1 (2) | 0 (0)
ESCHERICHIA INFECTION (Infections and infestations) | 0 (0) | 1 (1)
ESCHERICHIA SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
GASTROENTERITIS SALMONELLA (Infections and infestations) | 1 (1) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 3 (3) | 0 (0)
HERPES ZOSTER CUTANEOUS DISSEMINATED (Infections and infestations) | 1 (1) | 0 (0)
IMPETIGO (Infections and infestations) | 0 (0) | 1 (1)
INFECTED SKIN ULCER (Infections and infestations) | 1 (2) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 1 (1)
KLEBSIELLA BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0)
KLEBSIELLA SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (3) | 2 (3)
METAPNEUMOVIRUS INFECTION (Infections and infestations) | 1 (1) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 0 (0)
NEUTROPENIC SEPSIS (Infections and infestations) | 1 (1) | 1 (2)
OSTEOMYELITIS (Infections and infestations) | 0 (0) | 1 (1)
PARAINFLUENZAE VIRUS INFECTION (Infections and infestations) | 0 (0) | 1 (1)
PNEUMOCYSTIS JIROVECII INFECTION (Infections and infestations) | 1 (1) | 0 (0)
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 2 (2) | 0 (0)
PNEUMONIA (Infections and infestations) | 14 (15) | 8 (9)
PNEUMONIA FUNGAL (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA RESPIRATORY SYNCYTIAL VIRAL (Infections and infestations) | 1 (1) | 0 (0)
POST PROCEDURAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
PSEUDOMONAS INFECTION (Infections and infestations) | 0 (0) | 1 (1)
PULMONARY MYCOSIS (Infections and infestations) | 1 (1) | 0 (0)
PULMONARY SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 1 (1) | 0 (0)
RHINOVIRUS INFECTION (Infections and infestations) | 1 (1) | 0 (0)
SCROTAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
SCROTAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 2 (2) | 1 (1)
SEPTIC SHOCK (Infections and infestations) | 1 (1) | 0 (0)
SINUSITIS (Infections and infestations) | 0 (0) | 1 (1)
SOFT TISSUE INFECTION (Infections and infestations) | 1 (1) | 0 (0)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 (1) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 3 (3) | 0 (0)
UROSEPSIS (Infections and infestations) | 2 (2) | 0 (0)
VASCULAR DEVICE INFECTION (Infections and infestations) | 0 (0) | 1 (1)
VIRAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
ANASTOMOTIC LEAK (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 1 (1)
BLOOD GLUCOSE FLUCTUATION (Investigations) | 0 (0) | 1 (1)
CANDIDA TEST POSITIVE (Investigations) | 1 (1) | 0 (0)
ESCHERICHIA TEST POSITIVE (Investigations) | 1 (1) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 1 (1) | 0 (0)
CACHEXIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL DISORDER (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ACOUSTIC NEUROMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
BRONCHIAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CENTRAL NERVOUS SYSTEM LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CHRONIC LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
COLORECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
MALIGNANT NEOPLASM OF UNKNOWN PRIMARY SITE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 18 (18) | 4 (4)
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
PLASMA CELL MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
UTERINE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
ATAXIA (Nervous system disorders) | 1 (1) | 0 (0)
CEREBRAL INFARCTION (Nervous system disorders) | 1 (1) | 0 (0)
CHRONIC INFLAMMATORY DEMYELINATING POLYRADICULONEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0)
DISTURBANCE IN ATTENTION (Nervous system disorders) | 1 (1) | 0 (0)
HAEMORRHAGIC STROKE (Nervous system disorders) | 1 (1) | 0 (0)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0)
PROGRESSIVE SUPRANUCLEAR PALSY (Nervous system disorders) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 3 (3) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 (1) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1) | 0 (0)
DISORIENTATION (Psychiatric disorders) | 0 (0) | 1 (1)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 1 (1)
BLADDER DISORDER (Renal and urinary disorders) | 1 (1) | 0 (0)
CYSTITIS NONINFECTIVE (Renal and urinary disorders) | 1 (1) | 0 (0)
DYSURIA (Renal and urinary disorders) | 1 (1) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 1 (1)
VAGINAL PROLAPSE (Reproductive system and breast disorders) | 0 (0) | 1 (1)
BRONCHITIS CHRONIC (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
ERYTHEMA NODOSUM (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SKIN HAEMORRHAGE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
CIRCULATORY COLLAPSE (Vascular disorders) | 0 (0) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 (2) | 0 (0)
HYPERTENSIVE CRISIS (Vascular disorders) | 1 (1) | 1 (1)
HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Cohort (N=107) | Safety Expansion Cohort (N=51)
ANAEMIA (Blood and lymphatic system disorders) | 27 (55) | 11 (16)
AUTOIMMUNE HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 3 (4)
LEUKOPENIA (Blood and lymphatic system disorders) | 9 (14) | 2 (2)
NEUTROPENIA (Blood and lymphatic system disorders) | 47 (127) | 22 (49)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 24 (55) | 9 (20)
VERTIGO (Ear and labyrinth disorders) | 8 (9) | 2 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 8 (9) | 8 (9)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 4 (5) | 4 (4)
CONSTIPATION (Gastrointestinal disorders) | 11 (15) | 9 (10)
DIARRHOEA (Gastrointestinal disorders) | 42 (60) | 26 (45)
DYSPEPSIA (Gastrointestinal disorders) | 6 (6) | 3 (3)
FLATULENCE (Gastrointestinal disorders) | 4 (4) | 3 (4)
NAUSEA (Gastrointestinal disorders) | 35 (45) | 24 (32)
VOMITING (Gastrointestinal disorders) | 17 (21) | 2 (2)
CHILLS (General disorders) | 9 (9) | 5 (9)
FATIGUE (General disorders) | 27 (32) | 16 (18)
OEDEMA PERIPHERAL (General disorders) | 12 (15) | 5 (5)
PAIN (General disorders) | 9 (10) | 4 (5)
PYREXIA (General disorders) | 16 (22) | 6 (11)
BRONCHITIS (Infections and infestations) | 13 (17) | 0 (0)
CONJUNCTIVITIS (Infections and infestations) | 6 (7) | 3 (5)
HERPES ZOSTER (Infections and infestations) | 6 (7) | 5 (5)
INFLUENZA (Infections and infestations) | 6 (7) | 3 (3)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 (7) | 4 (6)
NASOPHARYNGITIS (Infections and infestations) | 19 (32) | 8 (11)
PNEUMONIA (Infections and infestations) | 7 (8) | 6 (6)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 11 (15) | 0 (0)
SINUSITIS (Infections and infestations) | 6 (7) | 4 (6)
SKIN INFECTION (Infections and infestations) | 0 (0) | 3 (4)
TOOTH INFECTION (Infections and infestations) | 2 (2) | 3 (3)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 22 (36) | 15 (20)
URINARY TRACT INFECTION (Infections and infestations) | 12 (15) | 8 (14)
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
FALL (Injury, poisoning and procedural complications) | 7 (8) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 8 (11) | 2 (3)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 6 (6) | 3 (3)
NEUTROPHIL COUNT DECREASED (Investigations) | 3 (6) | 3 (3)
PLATELET COUNT DECREASED (Investigations) | 3 (3) | 3 (5)
WEIGHT DECREASED (Investigations) | 6 (10) | 0 (0)
WEIGHT INCREASED (Investigations) | 7 (9) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 6 (6) | 1 (1)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 6 (9) | 6 (9)
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 17 (20) | 3 (4)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 14 (25) | 5 (6)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 3 (3) | 3 (5)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 4 (7) | 4 (6)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 10 (11) | 9 (12)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 13 (16) | 7 (8)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5)
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 9 (10)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 6 (10) | 4 (5)
DIZZINESS (Nervous system disorders) | 6 (7) | 7 (8)
HEADACHE (Nervous system disorders) | 16 (20) | 12 (12)
INSOMNIA (Psychiatric disorders) | 4 (4) | 4 (4)
POLLAKIURIA (Renal and urinary disorders) | 1 (1) | 3 (3)
COUGH (Respiratory, thoracic and mediastinal disorders) | 16 (20) | 14 (19)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 7 (10)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 2 (2)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (6)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 3 (3)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4)
UPPER-AIRWAY COUGH SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
ALOPECIA (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (4)
DRY SKIN (Skin and subcutaneous tissue disorders) | 7 (7) | 4 (5)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
PRURITUS (Skin and subcutaneous tissue disorders) | 7 (10) | 4 (4)
RASH (Skin and subcutaneous tissue disorders) | 11 (13) | 6 (6)
SKIN LESION (Skin and subcutaneous tissue disorders) | 2 (3) | 4 (4)
HYPERTENSION (Vascular disorders) | 15 (19) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2017-02-28): https://cdn.clinicaltrials.gov/large-docs/86/NCT01889186/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-27): https://cdn.clinicaltrials.gov/large-docs/86/NCT01889186/SAP_001.pdf